CLINICAL TRIAL: NCT02517450
Title: Effectiveness of an Adventure-based Training Programme in Promoting the Psychological Well-being of Primary School Children
Brief Title: Effectiveness of an Adventure-based Training Programme
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: UW 12-237
Record Dates: First submitted 2015-07-28; First posted 2015-08-07 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Healthy
Keywords: Subjects

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- experimental group (Experimental): The subjects had to participate an adventure-based training programme.
  Interventions: Behavioral: an adventure-based training programme
- placebo control group (Placebo Comparator): The subjects had to participate a placebo control programme
  Interventions: Other: a placebo control programme

INTERVENTIONS:
Behavioral: an adventure-based training programme — The programme consisted of five education sessions (around 75 minutes each) and a day's adventure-based training camp at the end of the academic year
  Arms: experimental group
Other: a placebo control programme — Subjects in the control group were invited to attend five 75-minute sessions of leisure activities, organised by a community centre, which included a cartoon film show, handicraft workshops, a health talk on the prevention of influenza and age-appropriate physical leisure activities, such as table tennis, badminton, chess and Chinese billiards. Additionally, they were invited to join a day visit to Hong Kong Ocean Park at the end of the academic year.
  Arms: placebo control group

SUMMARY:
This study tested the effectiveness of an adventure-based training programme in promoting the psychological well-being of primary schoolchildren. A randomised controlled trial was conducted, with 56 primary school pupils randomly assigned to the experimental group participating in the adventure-based training programme and 64 to the attention placebo control group.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong Chinese primary pupils from forms 5 and 6 of two schools were invited to participate in the study.

Exclusion Criteria:

* those with a chronic illness or identified cognitive and learning problems were excluded.

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2010-04; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
The Center for Epidemiologic Studies Depression Scale for Children at baseline | baseline
  baseline depressive symptoms
change of The Center for Epidemiologic Studies Depression Scale for Children at 9 months from baseline | 9 months
  depressive symptoms after the last intervention session
change of The Center for Epidemiologic Studies Depression Scale for Children at 12 months from baseline | 12 months
  depressive symptoms after 3 months from the last intervention session

SECONDARY OUTCOMES:
The Chinese version of the State Anxiety Scale for Children at baseline | baseline
  baseline anxiety level
change of The Chinese version of the State Anxiety Scale for Children at 9 months from baseline | 9 months
  anxiety level after the last intervention session
change of The Chinese version of the State Anxiety Scale for Children at 12 months from baseline | 12 months
  anxiety level after 3 months from the last intervention session
The Rosenberg Self-esteem Scale at baseline | baseline
  baseline self-esteem
change of The Rosenberg Self-esteem Scale at 9 month from baseline | 9 months
  self-esteem after the last intervention session
change of The Rosenberg Self-esteem Scale at 12 month from baseline | 12 months
  self-esteem after 3 months from the last intervention session
The Pediatric Quality of Life Inventory Generic at baseline | baseline
  baseline quality of life
change of The Pediatric Quality of Life Inventory Generic at 9 months from baseline | 9 months
  quality of life after the last intervention session
change of The Pediatric Quality of Life Inventory Generic at 12 months from baseline | 12 months
  quality of life after 3 months from the last intervention session

CONTACTS AND LOCATIONS:
Overall Officials: William, Ho Cheung LI, PhD, Principal Investigator — School of Nursing, The University of Hong Kong